CLINICAL TRIAL: NCT03814980
Title: A Home-based Intervention to Promote Mindful Breathing Awareness Through Pursed-lip Breathing Training for COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, M.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-004445
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: COPD; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Study (Experimental): Participants will be shown how to use a mindful breathing software application. The software will be used for 1 week. At the end of the week, participants will evaluate the software.
  Interventions: Behavioral: mindful breathing application; Device: application on a computer tablet

INTERVENTIONS:
Behavioral: mindful breathing application — Participants will use a mindful breathing application on a computer tablet.
Device: application on a computer tablet — a computer tablet

SUMMARY:
In this study, a system will be developed to guide patients with chronic obstructive pulmonary disease (COPD) to complete a mindful breathing practice at home. COPD is the third leading cause of death in the United States and no cure exists. Shortness of breath is the most common disabling symptom. Pursed lips breathing is a type of breathing practice that has demonstrated effectiveness for patients with COPD. It requires practice to maintain and there is currently no home system to provide the needed feedback and support to maintain PLB. Additionally, syncing breathing and heart rate variation offers patients additional benefits. The proposed project explores the use of biofeedback to guide COPD patients in a breathing practice and to provide data for health coaching to monitor and support the practice.

ELIGIBILITY:
Patients eligible for Pulmonary Rehabilitation will be recruited for this study.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of a mindful breathing application for COPD patients | About 1 week
  Mindful Breathing Application on a computer tablet for COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials